CLINICAL TRIAL: NCT05413720
Title: Study of the Innate Immune Response to the Acute Phase of Human Leptospirosis - IMMUNOLEPTO
Acronym: IMMUNOLEPTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017/CHU/14
Record Dates: First submitted 2022-06-03; First posted 2022-06-10 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-08

CONDITIONS: Leptospirosis
MeSH Terms: conditions — Leptospirosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with leptospirosis (Other)
  Interventions: Other: two additional blood samples specific to research

INTERVENTIONS:
Other: two additional blood samples specific to research — proportion of activated monocyte cells (CD14+CD16+ phenotype) within monocytes in the acute phase

SUMMARY:
The research hypothesis is based on a suspected strong involvement of the immune system in the genesis of serious manifestations of the disease (hepatitis, renal failure, thrombocytopenia, intra-alveolar hemorrhage). The question asked is that of the state of the immune system (quantitative and qualitative: activation markers, production of cytokines) evaluated by the study of circulating innate immune cells (monocytes, neutrophils, dendritic cells, lymphocytes, platelets).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 4 years;
* Weight ≥ 11 kg;
* with ongoing symptoms compatible with a clinical diagnosis of leptospirosis.
* AND having a diagnosis of leptospirosis confirmed according to standard care procedures: preferably by Polymerase Chain Reaction (PCR) (blood or urine) or, failing that, serology indicating a recent infection (positive Immunoglobulin M (IgM) or Microscopic Agglutination Test (MAT) technique with titer >1/400 for a pathogenic serogroup)
* AND affiliated to a Social Security scheme

Exclusion Criteria:

* Refusal of participation by the patient or his entourage if the patient is physically unable to give his opinion (coma, resuscitation, etc.).
* Not affiliated with social security
* Immunosuppression that may interfere with the interpretation of the results: chemotherapy in progress, immunosuppressants in progress for organ transplantation or autoimmune disease
* Patient under legal protection (Guardianship, Curators)

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
proportion of activated monocyte cells (CD14+CD16+ phenotype) within monocytes | at inclusion

CONTACTS AND LOCATIONS:
Locations (4):
- Reunion (4):
  - GHER, Saint-Benoît
  - CHU de la Réunion, Saint-Denis
  - CHOR, Saint-Paul
  - CHU de la Réunion, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No